CLINICAL TRIAL: NCT06368427
Title: A Non-interventional, Multi-centre Study to Investigate the Change in Patient-reported Outcomes in Moderate to Severe COPD Patients Newly Initiated on TRIXEO AEROSPHERE (Budesonide/Glycopyrronium/Formoterol) in Real-life Setting in Romania
Brief Title: Change in Patient-repOrted Outcomes in COPD Patients Newly Initiated on TRIXEO AEROSPHERE in Real worlD
Acronym: COnCORD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00100
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Glycopyrrolate; Formoterol Fumarate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients who initiate treatment with BGF MDI.: Patients with COPD, who are eligible for BGF MDI triple therapy. Patients are assigned to a therapeutic strategy within current routine care and not according to a clinical trial protocol. Every medical decision including the course of treatment will reflect exclusively the decision of the treating physician in a routine clinical situation according to the Summary of Product Characteristics of the corresponding medicinal products. There are no dose regimens or diagnostic procedures pre-defined.
  Interventions: Drug: budesonide / glycopyrronium / formoterol

INTERVENTIONS:
Drug: budesonide / glycopyrronium / formoterol — Trixeo Aerosphere 5 micrograms/7.2 micrograms/160 micrograms pressurised inhalation, suspension.
  The COnCORD study is an observational study that will be conducted in a real-life setting in Romania and is not designed to evaluate medicinal products given according to a specific randomised schedule. Treatment with BGF MDI treatment prescribed as per current practice, according to the SmPC and local market reimbursement criteria

SUMMARY:
The purpose of this study is to describe patients' clinical and self-reported outcomes of treatment with budesonide / glycopyrronium / formoterol Metered dose inhaler (BGF MDI) in Romania in real-life setting, up to 6 month of observation period. The study will focus primarily on the change in self-perceived health status in the first 12 weeks (3 months) of treatment with no pre-defined hypothesis.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, multi-centre study to investigate the change in patient-reported outcomes in moderate to severe COPD patients newly initiated on TRIXEO AEROSPHERE (budesonide / glycopyrronium / formoterol) in real-life setting in Romania. Furthermore, the patient satisfaction with the medication taken shall be assessed in the real-world setting; an important component that is not usually captured by RCTs. Patients with moderate to severe COPD who are eligible for BGF MDI therapy may be enrolled by physicians in the specialist care setting and the decision to prescribe BGF MDI must be independent of enrollment into the study.

This is a combined primary and secondary data collection study conducted to characterize the population of patients with COPD initiating triple therapy with BGF MDI in real-life setting. Thus, exposure data collected in this study will be primarily on BGF MDI treatment indicated for moderate to severe COPD patients as part of routine medical care. Primary data collection includes PROs; all other data will be documented based on the existing medical records (secondary data collection), either historically or throughout the period of 6-month follow-up, as part of the routine practical care of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed COPD
* Initiated treatment with BGF MDI as prescribed according to the summary of product characteristics (SmPC) and local market reimbursement criteria;
* Patients must be able and willing to read and to comprehend written instructions, and to comprehend and complete the questionnaires required by the protocol
* After full explanation, patients must have signed an informed consent document indicating that they understand the purpose of, and the procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* COPD due to known α-1 antitrypsin deficiency
* Previous treatment with triple fixed-dose combination in 12 months prior to baseline
* Hospitalization due to COPD exacerbation within the last 30 days prior to index date
* Pregnancy or lactation period
* Other uncontrolled disease, that might, in the investigator's opinion, influence the assessment for the current study
* Participation in a non-interventional, observational trial that might, in the investigator's opinion, influence the assessment for the current study, or participation in any interventional clinical trial in the last 30 days prior to baseline.
* Hospitalization for Covid-19 infection in the last 30 days prior to index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe COPD who are eligible for BGF MDI therapy may be enrolled by physicians in the specialist care setting.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 12 weeks (3 months) in the COPD Assessment Test (CAT) score | 12 weeks
  Compare COPD health status at baseline vs. 12 weeks of initiating treatment with BGF MDI

SECONDARY OUTCOMES:
Change from baseline to 6 months in the CAT score | 6 months
  Compare COPD health status at baseline vs. 6 months of initiating treatment with BGF MDI
Treatment Satisfaction Questionnaire for Medication (TSQM) scores after 12 weeks and 6 months of treatment | 6 months
  Evaluate treatment satisfaction after 12 weeks and 6 months of initiating treatment with BGF MDI
Percent responders of the CAT [MID=2] after 12 weeks of treatment | 12 weeks
  Describe frequency of Responder Rate based on the CAT after 12 weeks of initiating treatment with BGF MDI
Proportion of days covered (PDC) Time to discontinuation Reasons for treatment discontinuation | 6 months
  Describe patterns of BGF MDI usage including duration of therapy and discontinuation and reasons for discontinuation
Drivers for initiation or switch to BGF MDI via physician questionnaire | Baseline
  To describe the physicians' drivers for initiation or switch to BGF MDI

CONTACTS AND LOCATIONS:
Locations (16):
- Romania (16):
  - Research Site, Baia Mare
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Craiova
  - Research Site, Deva
  - Research Site, Dorohoi
  - Research Site, Hunedoara
  - Research Site, Iași
  - Research Site, Luduş
  - Research Site, Medgidia
  - Research Site, Oradea
  - Research Site, Sighișoara
  - Research Site, Suceava
  - Research Site, Târgu Mureş
  - Research Site, Timișoara

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/